CLINICAL TRIAL: NCT02635386
Title: Comparison of Dapagliflozin (DAPA) and Once-weekly Exenatide (EQW), Co-administered or Alone, DAPA/ Glucophage (DAPA/MET ER) and Phentermine/Topiramate (PHEN/TPM) ER on Metabolic Profiles and Body Composition in Obese PCOS Women
Brief Title: EQW, DAPA, EQW/DAPA, DAPA/MET ER and PHEN/TPM ER in Obese Women With PolycysticOvary Syndrome (PCOS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Woman's (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Karen Elkind-Hirsch, Director of Research, Woman's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP15-008; AZ ESR-14-10725 (Other Grant/Funding Number: Astra Zeneca,L.P)
Record Dates: First submitted 2015-12-15; First posted 2015-12-18 (Estimated); Results first posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Polycystic Ovary Syndrome; Obesity
Keywords: PCOS; GLP1 agonists; SGLT2 inhibitors
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity | interventions — Exenatide; Glucagon-Like Peptide 1; dapagliflozin; Sodium-Glucose Transporter 2 Inhibitors; Metformin; Qsymia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Exenatide once weekly (EQW ) (Experimental): EQW- 2 mg subcutaneous (SC) injection once every seven days for 24 weeks
  Interventions: Drug: Exenatide once weekly (EQW )
- Dapagliflozin (DAPA) (Experimental): DAPA-10 mg oral pill once daily in am for 24 weeks
  Interventions: Drug: Dapagliflozin (DAPA)
- EQW plus DAPA (Experimental): EQW- 2 mg SC injection once every seven days for 24 weeks DAPA-10 mg oral pill once daily in am daily for 24 weeks
  Interventions: Drug: EQW plus DAPA
- Dapagliflozin plus Glucophage (MET ER) (Experimental): Combination DAPA / MET ER-10 mg /2000 mg oral pill daily with food for 24 weeks
  Interventions: Drug: Dapagliflozin plus Glucophage (MET ER)
- Phentermine /Topiramate (PHEN/ TPM) ER (Active Comparator): Combination Phentermine /Topiramate ER -7.5 mg/46mg pill once daily in am for 24 weeks
  Interventions: Drug: Phentermine /Topiramate (PHEN/ TPM) ER

INTERVENTIONS:
Drug: Exenatide once weekly (EQW ) — 2 mg SC injection every 7 days
  Other Names: • Bydureon; • Long acting glucagon like peptide 1 (GLP1) agonist
  Arms: Exenatide once weekly (EQW )
Drug: Dapagliflozin (DAPA) — One pill (10 mg) by mouth daily (QD) in am
  Other Names: • Farxiga; • SGLT2 inhibitor
  Arms: Dapagliflozin (DAPA)
Drug: EQW plus DAPA — 2 mg SC injection every 7 days One pill (10 mg) by mouth QD in am
  Other Names: Bydureon plus Farxiga; Long acting GLP1 agonist plus SGLT2 inhibitor
  Arms: EQW plus DAPA
Drug: Dapagliflozin plus Glucophage (MET ER) — DAPA/MET ER-5 mg /1000 mg - 1 pill by mouth in am with food for 4 weeks DAPA/MET ER-10 mg /2000 mg - 2 pills in am by mouth with food -final dose
  Other Names: Xigduo; •Combination SGLT2 inhibitor and metformin ER
  Arms: Dapagliflozin plus Glucophage (MET ER)
Drug: Phentermine /Topiramate (PHEN/ TPM) ER — PHEN 3.75/TPM ER 23mg - 1 pill by mouth once daily in am for 2 weeks. After 2 weeks, PHEN 7.5mg/TPM ER 46mg- 1 pill by mouth once daily in am
  Other Names: Qsymia
  Arms: Phentermine /Topiramate (PHEN/ TPM) ER

SUMMARY:
This is a randomized, single-blind, parallel 5 treatment group 24-week trial designed to directly compare the therapeutic effects of exenatide once weekly (EQW), dapagliflozin (DAPA), EQW plus DAPA, combined DAPA/metformin extended release (XR) and the weight loss medication, phentermine/topiramate extended release (PHEN/TPM ER) on metabolic and endocrinological parameters in overweight/obese non-diabetic women with PCOS. In this study, we will examine the efficacy of these therapies on metabolic parameters, body weight and body composition, anthropometric measurements, and reproductive function in a well-defined group of pre-menopausal overweight/obese, non-diabetic women with PCOS, focusing on their relationship to insulin resistance and obesity. We hope to determine which treatment(s) addressing the multifaceted disturbances of individual subgroups emerge as the preferable therapy.

DETAILED DESCRIPTION:
Polycystic ovary syndrome is a heterogeneous condition characterized by disordered reproductive and metabolic function which accounts for the myriad of clinical features including androgen excess, chronic anovulation, insulin resistance adiposity, and dyslipidemia. This syndrome is highly prevalent, affecting between 8 and 18% of the female population, depending on the diagnostic criteria used. Hyperandrogenism, ovarian dysfunction and metabolic abnormalities - the main determinants of PCOS - all appear to be involved in a synergistic way in the pathophysiology of PCOS. Women with PCOS are more likely to be obese: between 38 and 88% of women with PCOS are overweight or obese, although PCOS can also manifest in lean women. Obesity, particularly abdominal obesity, plays a central role in the development of PCOS, and exacerbates the reproductive and metabolic dysfunction. Rather than absolute body weight, it is the distribution of fat that is important with central (visceral) adiposity being a risk factor. Visceral adipose tissue is more metabolically active than subcutaneous fat and the amount of visceral fat correlates with insulin resistance and hyperinsulinemia. Weight gain is also often an important pathogenic factor, with PCOS usually becoming clinically manifest in women with a presumable genetic predisposition for PCOS who subsequently gain weight. Therefore, environmental (particularly dietary) factors are important. However, BMI is also influenced by genetic factors such as the fat mass and obesity-associated protein, and obesity is a highly heritable condition. Therefore, the weight gain responsible for the manifestation of PCOS in many women with this condition is itself influenced by genetic factors. Ethnicity, genetic background, personal and family history, degree of obesity must all be taken into account because they might aggravate or even trigger metabolic disturbances women with PCOS. Moreover, the incidence of glucose intolerance, dyslipidemia, gestational diabetes, and type 2 diabetes (DM2) is increased in women with PCOS at all weight levels and at a young age. PCOS may be a more important risk factor than ethnicity or race for glucose intolerance in young women. The exact factors responsible for this excess risk in women with PCOS have not been identified; family history of DM 2, obesity, insulin resistance, beta cell (ß-cell) secretory dysfunction, and hyperandrogenism are possible candidates. With better understanding of its pathophysiology, the metabolic consequences of the syndrome are now evident. Therefore, these patients need to be followed up even after their presenting complaint has been adequately resolved.

Lifestyle modification is a key component for the improvement of reproductive function for overweight, anovulatory women with PCOS. Even a modest weight loss 5% of total body weight can restore ovulation in overweight women with PCOS. Features of PCOS (e.g., hirsutism, testosterone levels, insulin resistance, menstrual cyclicity and ovulation) showed marked improvements, and PCOS frequently resolved after substantial weight loss induced by bariatric surgery. Recently a number of anti-diabetes medications have been approved which facilitate weight loss and improve the underlying insulin resistance. We reported that treatment with the glucagon like peptide -1 (GLP-1) agonist, exenatide for 24 weeks was superior to single agent metformin treatment in improving insulin action and reducing body weight and hyperandrogenism in obese women with PCOS. We further observed exenatide treatment significantly improved first-phase insulin responses to oral glucose administration. Since aberrant first-phase insulin secretion and impaired suppression of endogenous glucose production are major contributors to postprandial hyperglycemia and development of type 2 diabetes, the effects of exenatide once weekly [EQW (2 mg)] to target these defects, and normalize glucose excursions are likely to be clinically significant in obese patients with PCOS. Sodium/glucose cotransporter 2 (SGLT-2) inhibitors are the newest class of medications for diabetes management that have not been investigated for use in the women with PCOS. The SGLT2 inhibitor, dapagliflozin [DAPA (10 mg/day)] has an insulin-independent action, promotes weight loss, has a low incidence of hypoglycemia, and complements the action of other antidiabetic agents. The loss of glucose with attendant caloric loss contributes to weight loss; in addition, improvements in β cell function have been seen. Because the SGLT2 inhibitors have a distinct mechanism of action that is independent of insulin secretion, the efficacy of this class of drugs is not anticipated to decline in the presence of severe insulin resistance. The weight loss seen with SGLT2 inhibitors is similar to that seen with glucagon-like peptide 1 agonists, and may be more acceptable because they are oral agents. The resulting weight loss will further assist in decreasing insulin resistance, leading to increased glucose disposal thus contributing to an increased insulin secretion-insulin sensitivity (ISSI) index, the primary outcomes measure.

The non-diabetic female with PCOS offers a unique model to study the relationship between insulin resistance and adiposity. Women with PCOS demonstrate abnormal body composition characterized by a greater percent body fat, body fat mass, and increased ratio of fat to lean mass (F/L ratio). Studies using dual-energy X-ray absorptiometry (DEXA) methodology report a higher degree of metabolic dysfunction in patients with PCOS which appears be directly associated with their higher F/L ratio. Given that monotherapy and combined therapy with exenatide once weekly (EQW),and dapagliflozin (DAPA) along with DAPA/ metformin XR therapy are associated with weight loss introduces a confounder to the current study since it prevents distinguishing direct effects of the compounds on β-cell function vs. effects due to reduced adiposity. To control for loss of body mass and provide appropriate intervention in the remaining study arm we propose the use of a comparator weight loss drug alone, combination phentermine (PHEN)/topiramate (TPM) extended release (ER). To avoid the confounding relationship of body fat and insulin resistance, we will enroll only obese non-diabetic women with PCOS. All patients will receive diet and lifestyle counselling, including advice on exercise, according to usual clinical routine commencing during the lead-in period and continuing throughout the study We propose a randomized, single-blind, parallel 5 treatment group 24-week trial designed to directly compare the therapeutic effects of exenatide once weekly (EQW), dapagliflozin (DAPA), EQW plus DAPA, combined DAPA/metformin ER and the weight loss medication, phentermine/topiramate extended release (PHEN/TPM ER) on metabolic and endocrinological parameters in obese non-diabetic women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

1. Non-diabetic women (18-45 years)
2. PCOS- NIH criteria hyperandrogenism and irregular menses
3. Obese class I, II, and III (BMI >30<45)
4. Willing to use effective contraception consistently during therapy which is defined as:

   1. an intrauterine device, tubal sterilization, or male partner vasectomy, or
   2. combination of two barrier methods with one being male condom.
5. Written consent for participation in the study

Exclusion Criteria:

1. Presence of significant systemic disease, heart problems including congestive heart failure, unstable angina or acute myocardial infarction, current infectious liver disease, acute stroke or transient ischemic attacks, history of pancreatitis, or diabetes mellitus (Type 1 or 2)
2. Any hepatic diseases in the past (infectious liver disease, viral hepatitis, toxic hepatic damage, jaundice of unknown etiology) or severe hepatic insufficiency and/or significant abnormal liver function tests defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN
3. Renal impairment (e.g., serum creatinine levels ≥1.4 mg/dL for women, or estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2) or history of unstable or rapidly progressing renal disease or end stage renal disease. Patients with a history of nephrolithiasis are also excluded due to increased association with kidney stone formation.
4. Uncontrolled thyroid disease (documented normal TSH), Cushing's syndrome, congenital adrenal hyperplasia or hyperprolactinemia
5. Significantly elevated triglyceride levels (fasting triglyceride > 400 mg/dL)
6. Untreated or poorly controlled hypertension (sitting blood pressure > 160/95 mm Hg)
7. Use of hormonal medications, lipid-lowering (statins, etc.), anti-obesity drugs or weight loss medications (prescription or OTC) and medications known to exacerbate glucose tolerance (such as isotretinoin, hormonal contraceptives, gonadotropin-releasing hormone agonists, glucocorticoids, anabolic steroids, C-19 progestins) stopped for at least 8 weeks. Use of anti-androgens that act peripherally to reduce hirsutism such as 5-alpha reductase inhibitors (finasteride, spironolactone, flutamide) stopped for at least 4 weeks
8. Prior history of a malignant disease requiring chemotherapy
9. Patients at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics should have careful monitoring of their volume status
10. History of unexplained microscopic or gross hematuria, or microscopic hematuria at visit 1, confirmed by a follow-up sample at next scheduled visit.
11. Presence of hypersensitivity to dapagliflozin or other SGLT2 inhibitors (e.g. anaphylaxis, angioedema, exfoliative skin conditions
12. Known hypersensitivity or contraindications to use GLP1 receptor agonists (exenatide, liraglutide)
13. Use of metformin, thiazolidinediones, GLP-1 receptor agonists, dipeptidyl peptidase 4 (DPP-4) inhibitors, SGLT2 inhibitors stopped for at least 4 weeks.
14. Prior use of medication to treat diabetes except gestational diabetes
15. Eating disorders (anorexia, bulimia) or gastrointestinal disorders
16. Suspected pregnancy (documented negative serum pregnancy test), desiring pregnancy in next 6 months, breastfeeding, or known pregnancy in last 2 months
17. Active or prior history of substance abuse (smoke or tobacco use within past 3 years) or significant intake of alcohol
18. Having a history of bariatric surgery
19. Patient not willing to use two barrier method contraception during study period (unless sterilized or have an IUD)
20. Patients with glaucoma or history of increased intraocular pressure, or use of any medications to treat increased intraocular pressure
21. Debilitating psychiatric disorder such as psychosis or neurological condition that might confound outcome variables. Patients with a history of bipolar disorder or psychosis, greater than one lifetime, episode of major depression, current depression of moderate or greater severity (PHQ-9score of 10 or more), presence or history of suicidal behavior or ideation with some intent to act on it, or antidepressant use that has not been stable for at least 3 months will also be excluded.
22. Inability or refusal to comply with protocol
23. Current participation or participation in an experimental drug study in previous three months

    -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Elkind-Hirsch, PhD, Principal Investigator — Woman's Hospital, Louisiana; Drake Bellanger, MD, Study Director — Woman's Hospital, Louisiana
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will only be shared with participant

REFERENCES:
- [Derived] Elkind-Hirsch KE, Chappell N, Seidemann E, Storment J, Bellanger D. Exenatide, Dapagliflozin, or Phentermine/Topiramate Differentially Affect Metabolic Profiles in Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2021 Sep 27;106(10):3019-3033. doi: 10.1210/clinem/dgab408. PMID 34097062

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 130 consented and 11 did not meet criteria and not randomized
Groups:
- Phentermine /Topiramate (PHEN/ TRP) ER: Combination Phentermine /Topiramate ER -7.5 mg/46mg pill once daily in am for 24 weeks
  Phentermine /Topiramate (PHEN/ TRP) ER: PHEN 3.75/TRP ER 23mg - 1 pill by mouth once daily in am for 2 weeks. After 2 weeks, PHEN 7.5mg/TRP ER 46mg- 1 pill by mouth once daily in am
Period: Overall Study
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TRP) ER
Started | 23 | 23 | 22 | 26 | 25
Completed | 20 | 17 | 20 | 19 | 16
Not Completed | 3 | 6 | 2 | 7 | 9
Not completed — Pregnancy | 2 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Moved Out of State | 0 | 1 | 0 | 0 | 0
Not completed — Noncompliant | 0 | 2 | 1 | 1 | 1
Not completed — side effects | 0 | 0 | 1 | 4 | 6
Not completed — needed other major surgery | 0 | 1 | 0 | 0 | 0
Not completed — Other medical problems not drug related | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants were started on medicine
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER | Total
Number analyzed (Participants) | 23 | 23 | 22 | 26 | 25 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (5.1) | 29.2 (6.3) | 31.4 (6.3) | 29.6 (7.0) | 29 (5.6) | 29.9 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 22 | 26 | 25 | 119
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 4 | 6 | 10 | 8 | 34
  White | 17 | 19 | 16 | 16 | 17 | 85
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 22 | 26 | 25 | 119
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — all patients were obese to enter trial
  kg/m^2 | 38.6 (5.1) | 38 (5.1) | 39.9 (4.2) | 37.6 (4.5) | 38.4 (4.4) | 38.3 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Oral Disposition (Insulin Sensitivity-insulin Secretion) Index
Description: An estimation of β-cell compensatory function, the insulin secretion-sensitivity index (IS-SI) will be derived by applying the concept of the oral disposition index to measurements obtained during the 2-h OGTT and calculated as the index of insulin secretion factored by insulin sensitivity (ΔINS/ΔPG 30 x Matsuda SIOGTT) from the OGTT. A higher score shows improved pancreatic insulin responsiveness relative to resistance.
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: index score
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
index score | 471 (83) | 311 (90) | 503 (80) | 395 (85) | 545 (93)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; Repeated Measure general linear model (SS/Drug treatments by visits) including arm of drug treatment as between subjects effect and visit (baseline and post 22-24 weeks treatment) as within subject effect; Test type: Superiority; p < 0.02, ANOVA; nested repeated measure

2. Secondary Outcome: Absolute Body Weight
Description: Treatment effect on body weight at 24 weeks of treatment
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: kilogram
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
kilogram | 100.4 (3.7) | 102.6 (4) | 99 (3.7) | 101.2 (3.8) | 97 (4.1)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Nested repeated measures design

3. Secondary Outcome: Body Mass Index (BMI)
Description: Treatment efficacy in reducing body mass at 24 weeks of treatment
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: kilogram/meter squared
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
kilogram/meter squared | 37.3 (1.1) | 37.4 (1.2) | 36.7 (1.1) | 37 (1.2) | 35.3 (1.3)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Nested repeated measures design

4. Secondary Outcome: Change in Percent Body Weight
Description: Treatment effect on change in percent body weight from baseline
Time Frame: Change from baseline (time 0) to study end (24 weeks)
Measure: Mean (Standard Error); unit: percentage change in body weight
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
percentage change in body weight | 3.8 (0.8) | 1.5 (1.4) | 6.9 (0.9) | 1.7 (1.0) | 8.1 (1.3)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; One way ANOVA with Bonferroni test to compare differences between groups if significant; Test type: Superiority; p < 0.0001, ANOVA; one way with Bonferroni contrast

5. Secondary Outcome: Central Adiposity (Waist Circumference)
Description: Treatment effect on loss of central adiposity after 24 weeks
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
centimeters | 104 (3) | 101 (3.2) | 106 (3) | 101.3 (3) | 97 (3.4)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Nested repeated measures design

6. Secondary Outcome: Waist-to-Hip Ratio (WHR)
Description: Treatment impact on central adiposity after 24 weeks
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
ratio | .83 (.016) | .79 (.017) | .86 (.016) | .83 (.016) | .81 (.018)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, ANOVA; Nested repeated measure design

7. Secondary Outcome: Waist-to-Height Ratio (WHtR)
Description: Treatment impact on WHtR which is a measure of central adiposity
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
ratio | .64 (.018) | .61 (.02) | .65 (.018) | .61 (.019) | .59 (.021)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Nested repeated measures design

8. Secondary Outcome: Total Fat Mass (kg) Evaluated by DEXA
Description: Treatment impact on total fat mass by DEXA
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: kilogram
Groups:
- Phentermine /Topiramate (PHEN/ TPM) ER: Combination Phentermine /Topiramate ER -7.5 mg/46mg pill once daily in am for 24 weeks
  Phentermine /Topiramate (PHEN/ TPM) ER: PHEN 3.75/TPMER 23mg - 1 pill by mouth once daily in am for 2 weeks. After 2 weeks, PHEN 7.5mg/TPM ER 46mg- 1 pill by mouth once daily in am
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
kilogram | 47.6 (2.4) | 47.8 (2.6) | 45.9 (2.4) | 48 (2.5) | 44.5 (2.8)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Nested repeated measures design

9. Secondary Outcome: Total Body Fat (%) by DEXA
Description: Treatment impact on percent total body fat by DEXA
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: percent fat mass
Groups:
- Phentermine /Topiramate (PHEN/ TPM) ER: Combination Phentermine /Topiramate ER -7.5 mg/46mg pill once daily in am for 24 weeks
  Phentermine /Topiramate (PHEN/ TPM) ER: PHEN 3.75/TPM ER 23mg - 1 pill by mouth once daily in am for 2 weeks. After 2 weeks, PHEN 7.5mg/TPMER 46mg- 1 pill by mouth once daily in am
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
percent fat mass | 46.1 (1.1) | 46.4 (1.2) | 45.8 (1.1) | 46.1 (1.1) | 45.2 (1.2)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Nested repeated measures design

10. Secondary Outcome: Android-Gynoid Ratio (AGR) as Determined by DEXA
Description: treatment impact on measure of central adiposity as determined by android/gynoid ratio
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
ratio | 1.07 (.024) | 1.02 (.03) | 1.04 (.02) | 1.04 (.03) | 1.03 (.03)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.01, ANOVA; Nested repeated measures design

11. Secondary Outcome: Trunk/Leg Fat Ratio by DEXA
Description: Treatment impact on trunk/limb ratio (measure of central adiposity) by DEXA
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
ratio | 1.03 (.045) | .95 (.048) | .93 (.045) | .98 (.047) | .99 (.05)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.035, ANOVA; Nested repeated measures design

12. Secondary Outcome: Fasting Blood Glucose
Description: Treatment impact on fasting concentration of glucose in the blood
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- Phentermine /Topiramate (PHEN/ TPM ER: Combination Phentermine /Topiramate ER -7.5 mg/46mg pill once daily in am for 24 weeks
  Phentermine /Topiramate (PHEN/ TPM) ER: PHEN 3.75/TPM ER 23mg - 1 pill by mouth once daily in am for 2 weeks. After 2 weeks, PHEN 7.5mg/TPM ER 46mg- 1 pill by mouth once daily in am
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
mg/dL | 91 (1.9) | 93 (2.1) | 86.5 (1.9) | 89 (2.0) | 91.4 (2.2)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Nested repeated measures design

13. Secondary Outcome: OGTT Mean Blood Glucose (MBG)
Description: Treatment effect on MBG measured during the oral glucose tolerance test
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
mg/dL | 118 (4.8) | 126.4 (5.2) | 112 (4.8) | 119 (4.9) | 113 (5.4)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.02, ANOVA; nested repeated measures design

14. Secondary Outcome: Fasting Insulin Sensitivity (HOMA-IR)
Description: Treatment effect on the ratio HOMA-IR which is insulin resistance measure derived from fasting blood glucose and insulin and is calculated by insulin (mU/ml)*glucose (mmol/L)/22,5. The higher thenumber the more insulin resistant.
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: index score
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
index score | 3.7 (0.55) | 3.6 (0.6) | 2.6 (0.55) | 3.3 (0.57) | 3.4 (0.62)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.035, ANOVA; Nested repeated measures design

15. Secondary Outcome: Matsuda Sensitivity Index Derived From the OGTT(SI OGTT)
Description: The SI IOGTT is a measure of peripheral insulin sensitivity derived from the values of Insulin (microunits per milliliter) and Glucose (milligrams per deciliter) obtained from the OGTT and the corresponding fasting values. SI (OGTT) = 10,000/ [(G fasting x I fasting) x (G OGTTmean x I OGTTmean)], where fasting glucose and insulin data are taken from time 0 of the OGTT and mean data represent the average glucose and insulin values obtained during the entire OGTT. The square root is used to correct for nonlinear distribution of insulin, and 10,000 is a scaling factor in the equation. The higher value, the more sensitive to insulin.
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: index score
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
index score | 3.1 (0.6) | 3.6 (0.7) | 3.9 (0.6) | 4.8 (0.6) | 4.7 (0.7)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Nested repeated measures design

16. Secondary Outcome: Corrected First Phase Insulin Secretion (IGI/HOMA-IR)
Description: Treatment effect on insulin secretion from 0 to 30 minutes after glucose load corrected for by fasting insulin sensitivity. A higher score shows improved first phase insulin secretion in response to glucose
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: index score
Groups:
- Phentermine /Topiramate (PHEN/ TPM) ER: Combination Phentermine /Topiramate ER -7.5 mg/46mg pill once daily in am for 24 weeks
  Phentermine /Topiramate (PHEN/ TPM ER: PHEN 3.75/TPM ER 23mg - 1 pill by mouth once daily in am for 2 weeks. After 2 weeks, PHEN 7.5mg/TPM ER 46mg- 1 pill by mouth once daily in am
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
index score | 1.03 (0.2) | 0.6 (0.21) | 0.91 (0.2) | 0.7 (0.2) | 1.1 (0.22)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.04, ANOVA; Nested repeated measures design

17. Secondary Outcome: Total Cholesterol Levels
Description: Treatment effect on blood concentrations of total cholesterol
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
mg/dL | 189 (10) | 186 (11) | 185 (10) | 192 (11) | 178 (12)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p > 0.05, ANOVA; Nested repeated measures design

18. Secondary Outcome: Triglyceride (TRG) Levels
Description: Treatment effect on blood concentrations of triglycerides
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
mg/dL | 130 (12) | 132 (13) | 112 (12) | 105 (12) | 110 (13)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.04, ANOVA; Nested repeated measures design

19. Secondary Outcome: Total Testosterone Concentrations
Description: Treatment effect on blood concentrations of total testosterone
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
ng/dL | 38.8 (4) | 35 (4.4) | 42.6 (4) | 39.5 (4.1) | 45.5 (4.5)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Nested repeated measures design

20. Secondary Outcome: Dehydroepiandrosterone Sulfate (DHEA-S) Levels
Description: Treatment effect on blood concentrations of DHEA-S
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: mcg/dL
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
mcg/dL | 165 (22) | 187 (24) | 169 (22) | 189 (23) | 201 (24)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, ANOVA; Nested repeated measures design

21. Secondary Outcome: Free Androgen Index (FAI)
Description: Treatment effect on FAI calculated from total testosterone divided by sex hormone binding globulin (SHBG) levels. A higher score indicates a worse outcome.
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: index score
Groups:
- Phentermine /Topiramate (PHEN/ TPM) ER: Combination Phentermine /Topiramate ER -7.5 mg/46mg pill once daily in am for 24 weeks
  Phentermine /Topiramate (PHEN/TPM) ER: PHEN 3.75/TPM ER 23mg - 1 pill by mouth once daily in am for 2 weeks. After 2 weeks, PHEN 7.5mg/TPM ER 46mg- 1 pill by mouth once daily in am
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
index score | 5.3 (0.72) | 4.7 (0.8) | 5.2 (0.73) | 5.7 (0.74) | 5 (0.8)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANOVA; Nested repeated measures design

22. Secondary Outcome: Systolic Blood Pressure (SBP)
Description: Treatment effect on SBP after 24 weeks of treatment
Time Frame: 24 weeks treatment
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
mmHg | 123.6 (1.9) | 123 (2.0) | 122 (1.9) | 128 (1.8) | 124 (2.0)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.035, ANOVA; Nested repeated measures design

23. Secondary Outcome: Diastolic Blood Pressure (DBP)
Description: Treatment effect on DBP after 24 weeks
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
Number analyzed (Participants) | 20 | 17 | 20 | 19 | 16
mmHg | 81 (1.7) | 79.8 (1.9) | 76 (1.7) | 82 (1.8) | 83.6 (2.0)
Statistical Analysis 1: Comparison: Exenatide Once Weekly (EQW ) vs Dapagliflozin (DAPA) vs EQW Plus DAPA vs Dapagliflozin Plus Glucophage (MET ER) vs Phentermine /Topiramate (PHEN/ TPM) ER; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.035, ANOVA; Nested repeated measures design

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Exenatide Once Weekly (EQW ) | Dapagliflozin (DAPA) | EQW Plus DAPA | Dapagliflozin Plus Glucophage (MET ER) | Phentermine /Topiramate (PHEN/ TPM) ER
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/22 | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/23 | 0/23 | 0/22 | 0/26 | 2/25
Other Adverse Events (participants affected / at risk) | 10/23 | 10/23 | 13/22 | 14/26 | 13/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (EQW ) (N=23) | Dapagliflozin (DAPA) (N=23) | EQW Plus DAPA (N=22) | Dapagliflozin Plus Glucophage (MET ER) (N=26) | Phentermine /Topiramate (PHEN/ TPM) ER (N=25)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0 | 2 — pregnancy was considered a serious AE and reported to the IRB, FDA and company
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (EQW ) (N=23) | Dapagliflozin (DAPA) (N=23) | EQW Plus DAPA (N=22) | Dapagliflozin Plus Glucophage (MET ER) (N=26) | Phentermine /Topiramate (PHEN/ TPM) ER (N=25)
Yeast infection or urinary tract infection (Renal and urinary disorders) | 0 | 6 | 7 | 7 | 0
Nausea and upset stomach (Gastrointestinal disorders) | 5 | 0 | 0 | 6 | 3
Injection site reaction (Skin and subcutaneous tissue disorders) | 5 | 0 | 4 | 0 | 0
Vaginal irritation (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Rapid heartbeat (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Insomnia (General disorders) | 0 | 0 | 0 | 0 | 3
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2
Lightheaded (General disorders) | 0 | 1 | 0 | 0 | 1
Headache (General disorders) | 0 | 0 | 0 | 0 | 2
Stuffy Nose (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Prolonged menstrual cycle (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Kidney Stone (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
One limitation of this study is the lack of a placebo only arm. As we were interested in the effects of different treatment regimens for obese women with PCOS, this study was designed to provide all patients with drug therapy. Limitations of the present study further include the absence of gold-standard measures of insulin sensitivity ; instead we used the OGTT using established surrogate measures.. Last, serial assessments were over only 24 weeks of treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT02635386/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2015-06-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT02635386/Prot_SAP_002.pdf